CLINICAL TRIAL: NCT06092632
Title: Efficacy of Pigmented Rice on Reducing Cardiometabolic Risk Factors Among Filipino Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Santo Tomas (Other)
Responsible Party: Principal Investigator, Diane S. Mendoza-Sarmiento, Principal Investigator, University of Santo Tomas
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: USantoTomas
Record Dates: First submitted 2023-10-10; First posted 2023-10-23 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Dyslipidemias; Overweight or Obesity; Hyperglycaemia (Non Diabetic)
Keywords: pigmented rice; dyslipidemia; hyperglycemia
MeSH Terms: conditions — Dyslipidemias; Overweight; Obesity; Hyperglycemia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pigmented Rice (Experimental): Cooked black pigmented rice will be consumed for six weeks (twice per day)
  Interventions: Other: Pigmented rice
- White Rice (Placebo Comparator): Cooked white rice will be consumed by the control group for six weeks (twice per day)
  Interventions: Other: White Rice

INTERVENTIONS:
Other: Pigmented rice — Cooked black rice
  Other Names: Black Rice
  Arms: Pigmented Rice
Other: White Rice — Cooked white rice
  Arms: White Rice

SUMMARY:
The primary purpose of this clinical trial is to investigate whether the consumption of pigmented rice (black rice) in the diet improves cardiovascular health, specifically body weight, lipids, and glucose levels. It also aims to know whether people enjoyed eating pigmented rice and if they would continue eating it.

DETAILED DESCRIPTION:
The goal of this clinical trial is to test if pigmented rice consumption can lower the cardiometabolic risk factors of adults. The main question[s] it aims to answer are:

* Will pigmented rice significantly reduce lipid levels compared to white rice after six weeks?
* Will pigmented rice significantly reduce glucose levels compared to white rice after six weeks? Will pigmented rice significantly reduce weight and waist-hip ratio levels compared to white rice after six weeks? What are the participants' experiences in consuming pigmented rice?

Participants will consume black-pigmented rice for six weeks while maintaining their usual physical activity. Researchers will compare the white rice group and the black rice group to see if lowers cardiometabolic risk factors.

ELIGIBILITY:
Inclusion Criteria:

* Aged 20-59 years.
* Body mass index between 18.5 -35 kg/m2
* Elevated cholesterol (total cholesterol >200 mg/dL or LDL cholesterol 130-190 mg/dL), and/or impaired fasting glucose (100-125mg/dL)
* Eat rice as a staple food at least twice per day

Exclusion Criteria:

* Are pregnant or lactating
* Regularly consume pigmented rice (two meals per day in the past 4 weeks)
* Have cardiovascular disease (hypertension, stroke, ischemic heart disease, myocardial infarction, or congestive heart failure) or diabetes mellitus
* Take cholesterol or glucose-lowering medications
* Have elevated blood pressure (>130/80 mmHg)
* Have an illness that may influence lipid metabolism or metabolic rate (liver cirrhosis, pancreatitis, chronic kidney disease, hyperthyroidism, hypothyroidism)
* Take supplements that may influence lipids and glucose levels (including polyphenols)
* Are on a strict diet regimen (calorie-restricted or excluding food groups, examples: (Examples: Ketogenic diet, Intermittent fasting, No Rice diet)
* Have an active lifestyle (Ex. Goes to the gym daily, regularly (≥3 times a week) and perform vigorous activities such as lifting weights, swimming, cycling fast or uphill, or running, or athlete)

Ages: 20 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-10-13 (Actual); Primary Completion 2024-08-30 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Change in Lipid Levels | six weeks
  Total cholesterol, Low-density lipoprotein, high-density lipoprotein, triglycerides
Change in Glucose Level | Six weeks
  Fasting blood glucose

SECONDARY OUTCOMES:
Change in Weight (kg) | Six weeks
  Weight in kilograms
Change in Waist Circumference (cm) | six weeks
  Waist circumference in centimeters
Change in Hip Circumference (cm) | Six weeks
  Hip Circumference in centimeters
Change in Waist:Hip (W:H ratio) | Six weeks
  Waist and hip measurement will be combined to report W:H ratio

CONTACTS AND LOCATIONS:
Overall Officials: Alison M Hill, Ph.D, Principal Investigator — University of South Australia; Elizabeth H Arenas, PhD, Principal Investigator — University of Santo Tomas
Locations (1):
- University of Santo Tomas, Manila, National Capital Region, Philippines

IPD SHARING:
Plan to Share IPD: No